CLINICAL TRIAL: NCT02535000
Title: Duloxetine as an Analgesic Agent in Patients Undergoing Elective Spine Surgery
Acronym: Duloxetine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Serviço de Anestesiologia de Joinville (Other)
Responsible Party: Principal Investigator, antonio bedin, MD, Serviço de Anestesiologia de Joinville
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 1
Record Dates: First submitted 2015-08-23; First posted 2015-08-28 (Estimated); Results first posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-09

CONDITIONS: Intervertebral Disc Degeneration
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group C (control) (Experimental): subjects who will receive one capsule of placebo before the surgery and being repeated the next day
  Interventions: Drug: Placebo
- Group D (duloxetine) (Active Comparator): subjects who will receive one capsule of duloxetine 60 mg before the surgery and being repeated the next day
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — duloxetine 60 mg
  Other Names: Cymbalta
  Arms: Group D (duloxetine)
Drug: Placebo — placebo
  Other Names: inactive substance
  Arms: Group C (control)

SUMMARY:
Duloxetine as an analgesic agent in patients undergoing elective spine surgery: evaluation with fentanyl demand controlled by the patient. The primary objective is to evaluate the efficacy of duloxetine in fentanyl consumption during the postoperative period of patients undergoing elective spine surgery by intervertebral disc degeneration . Secondary endpoints were pain scores and the presence or absence of adverse effects such as headache, nausea, vomiting, itching, dizziness and drowsiness.

DETAILED DESCRIPTION:
Multimodal analgesia is widely advocated for the control of perioperative pain in an attempt to reduce the use of opioids and their side effects. Duloxetine is a selective inhibitor of serotonin and norepinephrine reuptake with demonstrated efficacy in chronic pain such as painful diabetic neuropathy and postherpetic neuralgia. The primary objective is to evaluate the efficacy of duloxetine in fentanyl consumption during the postoperative period of patients undergoing elective spine surgery by intervertebral disc degeneration . Duloxetine as an analgesic agent in patients undergoing elective spine surgery: evaluation with fentanyl demand controlled by the patient. The primary objective is to evaluate the efficacy of duloxetine in fentanyl consumption during the postoperative period of patients undergoing elective spine surgery by degenerative disc disease. Secondary endpoints were pain scores and the presence or absence of adverse effects such as headache, nausea, vomiting, itching, dizziness and drowsiness.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included, of both genders, aged between 18 and 70 years and American Society of Anesthesiologists (ASA) physical status 1-3 and were eligible for the study

Exclusion Criteria:

* Patients allergics to duloxetine, ketoralac or fentanyl, pre-existing history of use of illegal substances or alcohol in an abusive manner and abnormal kidney or liver function tests.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-10-20 (Actual); Study Completion 2015-10-30 (Actual)

REFERENCES:
- [Result] Bedin A, Caldart Bedin RA, Vieira JE, Ashmawi HA. Duloxetine as an Analgesic Reduces Opioid Consumption After Spine Surgery: A Randomized, Double-Blind, Controlled Study. Clin J Pain. 2017 Oct;33(10):865-869. doi: 10.1097/AJP.0000000000000471. PMID 28002096

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was started in January, 2014 at the Centro Hospitalar Unimed of Joinville, Brazil
Period: Overall Study
Arm/Group | Group C (Control) | Group D (Duloxetine)
Started | 30 | 30
Completed | 29 | 28
Not Completed | 1 | 2
Not completed — Cancellation of surgery. | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group C (Control) | Group D (Duloxetine) | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 28 | 57
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 13 | 13 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Brazil | 29 | 28 | 57

OUTCOME MEASURES:

1. Primary Outcome: Total Consumption of Fentanyl (in Micrograms) Self-administered by the Patient and Accessed at 24 and 48 Hours After Spine Surgery.
Description: The main evaluation parameter was the total consumption of fentanyl (in micrograms) self-administered by the patient and accessed at 24 and 48 hours after surgery. At the beginning of the study, Group C (placebo) would have 30 patients and D (duloxetine) would also have 30 patients. However, 1 patient in Group C and 2 patients in Group D were excluded due to the cancellation of the proposed surgery, after the patient had received 60 milligrams of duloxetine. The lower the consumption of fentanyl, the better the analgesic effect of duloxetine.
Time Frame: up to 2 days.
Population: At the beginning of the trial, Group C would have 30 patients and D also 30 patients. However, 1 patient in Group C and 2 patients in group D were excluded due to cancellation of the proposed surgery, after patient receiving 60 mg of duloxetine. The lower the consumption of fentanyl, the better the analgesic effect of duloxetine.
Measure: Mean (Standard Deviation); unit: micrograms
Arm/Group | Group C (Control) | Group D (Duloxetine)
Number analyzed (Participants) | 29 | 28
micrograms
  Fentanyl consumption in between 0 and 24 hours. | 726 (36) | 503 (19)
  Fentanyl consumption in between 24 and 48 hours. | 180 (20) | 136 (13)

2. Secondary Outcome: Self Reported Pain Score Range From 0 (no Pain) to 10 (Worst Possible Pain).
Description: At the beginning of the study, Group C (placebo) would have 30 patients and D (duloxetine) would also have 30 patients. However, 1 patient in Group C and 2 patients in Group D were excluded due to the cancellation of the proposed surgery, after the patient had received 60 milligrams of duloxetine. Self reported pain score range from 0 (no pain) to 10 (worst possible pain) 2, 6, 12, 24, 36 and 48 hours after surgery. Higher scores mean a worse score and low scores mean a better score.
Time Frame: up to 2 days.
Population: At the beginning of the study, Group C (placebo) would have 30 patients and D (duloxetine) would also have 30 patients. However, 1 patient in Group C and 2 patients in Group D were excluded due to the cancellation of the proposed surgery, after the patient had received 60 milligrams of duloxetine.
Measure: Mean (Standard Deviation); unit: Number (pain score range 0 to 10).
Arm/Group | Group C (Control) | Group D (Duloxetine)
Number analyzed (Participants) | 29 | 28
Number (pain score range 0 to 10).
  Pain score 2 hours after surgery. | 2.27 (2.67) | 2.14 (2.04)
  pain score 6 hours after surgery | 2.67 (2.44) | 2.28 (2.07)
  Pain score 12 hours after surgery. | 2.10 (2.31) | 2.07 (1.92)
  Pain score 24 hours after surgery. | 1.68 (2.13) | 1.66 (1.64)
  Pain score 36 hours after surgery. | 1.48 (2.06) | 1.37 (1.52)
  Pain score 48 hours after surgery. | 1.51 (2.08) | 1.07 (1.03)

ADVERSE EVENTS:
Time Frame: Two days.
Description: Incidence of adverse effects accessed in the first two postoperative days.
Arm/Group | Group C (Control) | Group D (Duloxetine)
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 10/29 | 9/28
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group C (Control) (N=29) | Group D (Duloxetine) (N=28)
somnolence (Nervous system disorders) | 5 (5) | 4 (4)
itching (General disorders) | 2 (2) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
We used the same dose as previous investigators. We did not evaluate a possible effect of duloxetine on chronic postsurgical pain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No